CLINICAL TRIAL: NCT03828071
Title: National Clinical Research Center of Kidney Diseases, Jinling Hospital
Brief Title: Autologous Hematopoietic Stem Cell Transplantation for Refractory Lupus Nephritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, M.D., Director, Nanjing University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-1008
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- stem cell transplantation (Other): patients enrolled in this study will received autologous hematopoietic stem cell transplantation as the initial treatment.
  Interventions: Procedure: Autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Autologous hematopoietic stem cell transplantation — Stem cell mobilization and collection: Peripheral blood stem cells were mobilized with cyclophosphamide (2.0 g/m2) for 2 days and granulocyte colony-stimulating factor (G-CSF) at 5-10 μg/kg per day was administered when the level of peripheral leucocytes was < 1×109/L. Peripheral leukocyte counts were monitored, and harvesting was performed when the peripheral white blood cell level rebounded .
  Conditioning and reinfusion of stem cells: The conditioning regimen consisted of intravenous cyclophosphamide (40 mg/kg/day × 4 days) 5 days before transplantation (a total dose 160 mg/kg) and rabbit antithymocyte globulin (ATG) (2.5mg/kg/day × 3 days) 4 days before transplantation. The dose of cyclophosphamide and ATG could be reduced according to the patients' condition.

SUMMARY:
In this study, we aimed to evaluate the long term efficacy, remission, survival and safety of autologous hematopoietic stem cell transplantation in patients with refractory lupus nephritis.

This is an single arm, non-randomized study. Patients who were diagnosed with relapsed and refractory lupus nephritis would included in this study. Refractory lupus nephritis is defined as no response to at least one type of immunosuppressant therapy (including corticosteroids, cyclophosphamide, tacrolimus, mycophenolate mofetil and cyclosporine) for more than six months, or relapse during the period maintenance therapy with kidney pathological transformation or persistently positive antibodies. Close observation was carried out at stem cell harvest, at transplantation, at 3, 6, 12, 18, and 24 months and then once a year after autologous stem cell transplantation.

20-30 cases will be included in this study.

DETAILED DESCRIPTION:
Treatment plan: Peripheral blood stem cells were mobilized with cyclophosphamide (2.0 g/m2) for 2 days and granulocyte colony-stimulating factor (G-CSF) at 5-10 μg/kg per day was administered when the level of peripheral leucocytes was < 1×109/L. Peripheral leukocyte counts were monitored, and harvesting was performed when the peripheral white blood cell level rebounded (usually 11 days after cyclophosphamide). The target acquisition was CD34+ cells > 2×10^6/kg and mononuclear cells > 2×10^8/kg. The graft was preserved at a temperature of -196 ℃ for further use. The conditioning regimen consisted of intravenous cyclophosphamide (40 mg/kg/day × 4 days) 5 days before transplantation (a total dose 160 mg/kg) and rabbit antithymocyte globulin (ATG) (2.5mg/kg/day × 3 days) 4 days before transplantation. The dose of cyclophosphamide and ATG could be reduced according to the patients' condition. Methylprednisolone (80-500 mg/day) was administered through intravenous drip at the same time with ATG to reduce anaphylaxis. The incidence of drug-related complications was decreased by hyperhydration (the volume of infusion liquid is 50 ml/kg/day), urine alkalization (infusion of sodium bicarbonate 250ml/day), and anti-emetic medication. G-CSF (0.5 μg/kg/d) was administered to each patient beginning the day after stem cells reinfusion until the level of absolute peripheral neutrophil count was consecutively higher than 1.0 × 10^9/L.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed with relapsed and refractory lupus nephritis; 2. Ages from 14 - 45 years old; 3. Serum creatinine < 2mg/dl; 4. Alanine aminotransferase < 2 times of normal upper limit; 5. Left ventricular ejection fraction > 50%; 6. Subjects (or their legal representatives) must signed an informed consent document.

Exclusion Criteria:

* 1. Active infection; 2. Known or suspected hypersensitivity to CTX or ATG; 3. Subjects suffering from uncontrolled or severe cardiovascular disease; 4. Subjects suffering from serious physical disease and mental illnesses.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Renal remission rate | seven years
  The curative effect on the kidney was defined as follows: complete remission: proteinuria< 0.4 g/24 h, red blood cell (RBC) < 3/HP in urine sediment, serum albumin > 3.5g/dl and serum creatinine < 1.24 mg/dl; partial remission: 50% baseline < decrease of proteinuria < 3.5 g/24 h, serum albumin >30g/L and serum creatinine < 1.24 mg/dl, no remission (NR): failed to achieve partial remission

SECONDARY OUTCOMES:
renal survival | seven years
  the time from treatment start to dialysis.
treatment related mortality | 3 months
  patients who dies in 3 months after treatment start.

CONTACTS AND LOCATIONS:
Overall Officials: zhihong liu, MD, Principal Investigator — National Clinical Research Center of Kidney Diseases, Jinling Hospital
Locations (1):
- National Clinical Research Center of Kidney Diseases, Jinling Hospital, Nanjing, Jiangsu, China